CLINICAL TRIAL: NCT02439073
Title: Postoperative Rehabilitation in Operation for LUng CAncer (PROLUCA) - A Randomized Clinical Trial With Blinded Effect Evaluation
Brief Title: Postoperative Rehabilitation in Operation for LUng CAncer (PROLUCA)
Acronym: PROLUCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jesper Holst Pedersen, MD, MrDSci, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H-3-2012-028
Record Dates: First submitted 2015-01-29; First posted 2015-05-08 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early initiated rehabilitation (Experimental): A supervised 12-week rehabilitation program, initiated two weeks post surgery, containing 24 group-based exercise sessions, three individual counseling sessions, and three group-based lessons in health-promoting behavior. If the participants have special needs in terms of smoking cessation, nutritional counseling or patient education, this is offered too.
  Interventions: Behavioral: Rehabilitation
- late initiated rehabilitation (Active Comparator): A supervised 12-week rehabilitation program, initiated 14 weeks post surgery, containing 24 group-based exercise sessions, three individual counseling sessions, and three group-based lessons in health-promoting behavior. If the participants have special needs in terms of smoking cessation, nutritional counseling or patient education, this is offered too.
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation — The postoperative intervention are the same in both intervention groups and consists of a supervised 12-week rehabilitation program containing 24 group-based exercise sessions, three individual counseling sessions, and three group-based lessons in health-promoting behavior. If the participants have special needs in terms of smoking cessation, nutritional counseling or patient education, this is offered too.The postoperative physical exercise consists of an individually prepared supervised strength exercise - and a group-based cardiovascular exercise twice a week (60 minutes/session) on non-consecutive days for 12 weeks, a total of 24 sessions.
  Other Names: exercise intervention

SUMMARY:
Purpose The purpose of the PROLUCA study is to investigate the efficacy of early postoperative rehabilitation in a non-hospital setting in patients with operable lung cancer, with focus on exercise training.

Design/Methods

One hundred and twenty-eight (n=128) participants (64 patients/study arm) with Non-Small Cell Lung Cancer (NSCLC), stage I-IIIa, referred for surgery, will be randomized to one of the following two groups:

1. Early postoperative rehabilitation initiated as early as two weeks after surgery
2. Postoperative rehabilitation initiated 14 weeks after surgery Intervention The intervention consists of a supervised group exercise program comprising resistance and cardiorespiratory exercise two hours weekly for 12 weeks combined with individual counseling.

The primary study endpoint is Maximal oxygen uptake measured by a VO2peak test (direct measurement) Secondary endpoints include: Six minutes walk distance (6MWD), One-repetition-maximum (1RM) Patient-reported outcomes (PROs) on health related quality of life, fatigue, depression, lifestyle, postoperative complications, hospitalization time, sick leave, work status and survival.

Results The results of PROLUCA will identify the optimal timing of postoperative rehabilitation in NSCLC patients with focus on increasing physical capacity and health related quality of life and reducing the side effects from the treatment of the cancer disease.

ELIGIBILITY:
Inclusion Criteria:

* All subjects are assigned for curative lung cancer surgery at Department of Cardiothoracic Surgery RT at Copenhagen University Hospital (Rigshospitalet)
* Performance status 0-2 (WHO)
* Living in the City of Copenhagen or surrounding Municipalities
* Ability to read and understand Danish
* Approval by primary surgeon

Exclusion Criteria:

* Presence of metastatic disease or surgical inoperability. Diagnosis of Lung Cancer not verified by histological diagnosis.
* Decompensated heart failure, severe aortic stenosis, uncontrolled arrhythmia, acute coronary syndrome
* Contraindications to maximal exercise testing as recommended by the American Thoracic Society and exercise testing guidelines for cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2014-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
A change in maximum oxygen consumption | A change in maximum oxygen consumption from baseline to post intervention (for group one, the experimental group, it is approximately 14 weeks after the operation and for group two it is approximately 26 weeks after the operation)
  A change in maximum oxygen consumption from baseline to post interventon, measured by a VO2peak, evaluated by an incremental test using an electromagnetically braked cycle ergometer

SECONDARY OUTCOMES:
Patient Reported outcomes | Baseline, post intervention, follow-up at 26 and 52 weeks after surgery
  EORTC QLQ-C30, EORTC-LC13, FACT-L, SF-36, HADS, The distress thermometer, MSPSS, PAS2
Six minutes walk distance | Baseline, two and 8 weeks after surgery. post intervention, follow-up at 26 and 52 weeks after surgery
Lung capacity | Baseline, two and 8 weeks after surgery. post intervention, follow-up at 26 and 52 weeks after surgery
  Spirometry
Muscle strength chest and leg press | Baseline, post intervention, follow-up at 26 and 52 weeks after surgery
  one repetition maximum
A change in maximum oxygen consumption | A change in maximum oxygen consumption from baseline to 52 weeks after operation
  measured by a VO2peak, evaluated by an incremental test using an electromagnetically braked cycle ergometer

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H. Pedersen, MD, MrDSci, Study Director — Rigshospitalet, Denmark
Locations (1):
- Copenhagen Centre for Cancer and Health, Copenhagen, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided